CLINICAL TRIAL: NCT03392545
Title: Combination of Immunization and Radiotherapy for Malignant Gliomas (InSituVac1)
Acronym: InSituVac1
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Tiantan Hospital (Other)
Collaborators: Duke University (Other)
Responsible Party: Principal Investigator, Song Lin, MD and Chief Physician, Beijing Tiantan Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B0011
Record Dates: First submitted 2017-12-11; First posted 2018-01-08 (Actual); Last update posted 2019-07-11 (Actual); Status verified 2019-07

CONDITIONS: High Grade Glioma; Glioblastoma; Glioma of Brainstem; Glioma, Malignant
Keywords: gliomas; radiotherapy; immunetherapy
MeSH Terms: conditions — Glioma; Glioblastoma | interventions — Radiation; Granulocyte-Macrophage Colony-Stimulating Factor; Poly I-C

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Combined immune adjuvants and radiation (Experimental): Patients with malignant gliomas will receive combined immune adjuvants (GM-CSF, TLR ligands) and radiation. The safety and efficacy will be analyzed.
  Interventions: Combination Product: Combined immune adjuvants and radiation

INTERVENTIONS:
Combination Product: Combined immune adjuvants and radiation — 24 hours before the radiation, patients will be administrated poly I:C or CAR-T or TCR-T intratumorally and receive granulocyte macrophage colony stimulating factor 5 days after the radiation.
  Other Names: GM-CSF, poly I:C and radiation; CAR-T; TCR-T

SUMMARY:
The study will investigate combined radiotherapy and immunotherapy on malignant gliomas. Immune adjuvants will be injected intratumorally and systemically to induce antitumor-specific immunity after radiation induced immunological tumor cell death (ICD). With radiation, tumor cells release tumor antigens that are captured by antigen presenting dendritic cells. Immune adjuvants promote the presentation of tumor antigens and the priming of antitumor T lymphocytes. The combined treatment induces and amplifies the specific antitumor immunity in patients with malignant gliomas, prolonging survivals of patients.

DETAILED DESCRIPTION:
High grade gliomas, such as glioblatoma (GBM) is an aggressive malignancy with a poor prognosis. The current strategy for newly diagnosed GBM patients includes surgery, chemotherapy and radiotherapy. Unfortunately, after the standard treatmetn,the median survival of GBM is only about one year. Once relapsed, there is no standard therapy and survival is less than 9 months. Recently, personalized cancer immunotherapy has shown great promise in treating different types of cancers. However, effective immunotherapies for high grade gliomas, especially after progression, have yet to be established. Newly diagnosed GBM patients experience recurrence in five or seven months after standard treatment. We will investigate whether combining radiotherapy with intratumoral and systemic administration of immune adjuvants will improve the treatment outcome of high grade gliomas. We will use several immune adjuvants that activate innate and adaptive immunity.

ELIGIBILITY:
Inclusion Criteria:

1. Histopathologically confirmed glioma
2. Age18-65
3. Participants had undergone maximal surgical resection
4. Amount of dexamethasone was not more than 2mg/ days
5. Ability and willingness to sign informed consent
6. Karnofsky Performance Score of 70 or more
7. Normal liver and kidney function
8. Not accepted other treatment plan during the immunotherapy

Exclusion Criteria:

1. Not conforming to the standard
2. Systemic illness or medical condition may pose additional risk,including cardiac, incompensated renal or liver function abnormalities;inflammatory and immune system diseases of rheumatic arthritis
3. Received other drugs for glioma therapy 60days before participated
4. Allergy to immune adjuvant
5. Nervous system disease and diffuse leptomeningeal disease
6. Amount of dexamethasone was more than 2mg/days during the immunotherapy
7. Pregnant or lactation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-04-01 (Actual); Primary Completion 2020-04-01 (Estimated); Study Completion 2020-06-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-related Adverse Events | 2 years
  Adverse events during and after the combined treatment

SECONDARY OUTCOMES:
Progression-free Survival | 2 years
  Disease progression free survival time after combined treatment
Overall Survival | 2 years
  Overall survival time after the combined treatment

CONTACTS AND LOCATIONS:
Overall Officials: Peijuan Ren, M.D., Study Director — Beijing Tiantan Hospital; Song Lin, M.D., Principal Investigator — Beijing Tiantan Hospital; You-Wen He, M.D. Ph.D., Principal Investigator — Duke University
Locations (1):
- Beijing Tiantan Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Zheng Y, Jiang H, Yang N, Shen S, Huang D, Jia L, Ling J, Xu L, Li M, Yu K, Ren X, Cui Y, Lan X, Lin S, Lin X. Glioma-derived ANXA1 suppresses the immune response to TLR3 ligands by promoting an anti-inflammatory tumor microenvironment. Cell Mol Immunol. 2024 Jan;21(1):47-59. doi: 10.1038/s41423-023-01110-0. Epub 2023 Dec 4. PMID 38049523
- [Derived] Jiang H, Yu K, Cui Y, Ren X, Li M, Yang C, Zhao X, Zhu Q, Lin S. Combination of Immunotherapy and Radiotherapy for Recurrent Malignant Gliomas: Results From a Prospective Study. Front Immunol. 2021 May 7;12:632547. doi: 10.3389/fimmu.2021.632547. eCollection 2021. PMID 34025640